CLINICAL TRIAL: NCT05942105
Title: A Retrospective Multicentric Clinical Study Comparing Different Techniques for Intraoperative Localization of Non-palpable Breast Lesions During Breast Conservative Surgery
Brief Title: Different Localization Techniques for Non-palpable Breast Lesions Comparison: a Retrospective and Multicentric Clinical Study
Acronym: Localization01
Status: Active, not recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Fabio Corsi, Professor, Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: 2776
Record Dates: First submitted 2023-06-27; First posted 2023-07-12 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- ROLL technique: Radioguided occult lesion localization
  Interventions: Procedure: Breast conservative surgery
- MAGNETIC SEED: Magnetic seed localization
  Interventions: Procedure: Breast conservative surgery
- WGL technique: Wire guided localization for non-palpable breast lesions
  Interventions: Procedure: Breast conservative surgery
- CARBON: Carbon dye localization for non-palpable breast lesions
  Interventions: Procedure: Breast conservative surgery

INTERVENTIONS:
Procedure: Breast conservative surgery — Breast conservative surgery after non-palpable lesion localization

SUMMARY:
Breast conservative surgery (BCS) is nowadays the standard of care for patients affected by early breast lesions. Screening programmes led to an increase of non-palpable breast lesion detection rates. These patients are often eligible for BCS and an accurate preoperative localization technique for the detection of the lesion is required to guarantee a safe surgical excision. The primary goal of BCS is to obtain a complete resection of the tumor with disease-free surgical margins. The presence of tumor on surgical margins on postoperative histological examination of the specimen increases the risk of local recurrence and it requires a surgical re-excision. For all these reasons different techniques for localization of non-palpable breast lesions have been developed over time. Since '70s the wire guided localization (WGL) technique has represented the gold standard; however it has several limitations such as wire migration or fracture and patient referred discomfort related to wire placement. Over time, other techniques have been proposed, such as the radioguided occult lesion localization (ROLL), radioactive and magnetic seeds, carbon dye and ultrasound-guided preoperative localization.

Currently there are several studies of comparison between the WGL and the more modern techniques. All of these data claim the effectiveness of the new "wire-free" methodics ensuring a safe surgical resection with tumor-free margins and, in some cases, a better aesthetic result.

Studies of comparison between the modern techniques are limited. There is no scientific evidence of the superiority of a technique over the other. A multicentric Italian survey demonstrated that the most used localization techniques nowadays are the WGL, ROLL, the magnetic seed and the carbon dye.

The aim of this retrospective study is to compare these techniques to assess their efficacy in the localization of non-palpable breast lesions.

ELIGIBILITY:
Inclusion Criteria:

* Female sex;
* Patients who underwent breast conservative surgery for non-palpable occult breast lesions;
* Intraoperative localization of breast lesion with WGL, ROLL, magnetic seed, carbon dye;
* Preoperative diagnosis on histology or cytology of borderline lesion (B3 or C3) or malignant lesion (B4-B5 or C4-C5).

Exclusion Criteria:

* Diagnosis of benign breast lesion, both on preoperative needle breast biopsy (B2) or on fine needle breast aspiration (C2);
* Clinically palpable breast lesion;
* Localization of a non-palpable lesion through two or more different techniques;
* Breast tumor localization with clip in patients who underwent neoadjuvant chemotherapy.

Ages: 18 Years to 85 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients with non-palpable breast lesion candidated for conservative surgery
Sampling Method: Probability Sample
Enrollment: 1064 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Free-surgical margins | 6 months
  Number of surgical procedures in which surgical margins are disease-free ("no ink on tumor" for invasive cancer and margin of 2 mm for in situ-carcinoma)

SECONDARY OUTCOMES:
Excess breast resection | 6 months
  Excess breast resection calculated by the "calculated resection ratio" (CRR=total resection volume/optimal resection volume)
Surgery time | 6 months
  Surgery duration
Hospitalization days | 6 months
  Number of hospitalization days
Complications | 6 months
  Complications (after biopsy or surgery)
Reintervention | 6 months
  Reintervention rates
Follow up | 5 years after enrollment
  5-years follow-up outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Lombardy, Italy